CLINICAL TRIAL: NCT00594451
Title: Gene-Environment Interactions in RA Autoimmunity Disease Severity
Brief Title: Gene-Environment Interactions in Rheumatoid Arthritis Autoimmunity Disease Severity
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: University of Alabama at Birmingham (Other); University of Colorado, Denver (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0358-06-NH; 1R03AR054539-01 (NIH)
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; cigarette smoking; gene-environmental interactions; autoimmunity; disease severity
MeSH Terms: conditions — Arthritis, Rheumatoid; Cigarette Smoking; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — All subjects will provide baseline serum and DNA.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- I Multicenter Veteran's Affairs Rheumatoid Arthritis (VARA) registry: multicenter Veteran Affairs Rheumatoid Arthritis (VARA) registry
- II NIH-funded Consortium for the Longitudinal Evaluation of African Americans with Early RA (CLEAR): NIH-funded Consortium for the Longitudinal Evaluation of African Americans with Early RA (CLEAR)

SUMMARY:
The objective of the proposed study is to assess the role of smoking and complex gene-smoking interactions in two understudied Rheumatoid Arthritis (RA)groups.

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) is a systemic inflammatory disease affecting over 2 million people in the U.S. alone, a condition characterized by progressive joint destruction, significant work-related disability and accelerated mortality. While the precise cause of RA is unknown, it is clear that the disease does not result from a single heritable factor or single environmental exposure. Of the many environmental exposures that have been studied, cigarette smoking is the factor most consistently shown to be associated with RA onset. In addition to its role in disease susceptibility, recent studies have found that smoking, along with genetic factors, contribute to RA-related autoimmunity and disease severity. Moreover, studies to date looking at disease severity in RA have exclusively involved women of Caucasian/European ancestry. This is an important distinction since although RA is more common in women, smoking appears to be most closely linked to RA risk in men. Additionally, the burden of other smoking-related illnesses appears to be greatest among non-Caucasian populations. For this reason and because smoking rates and prevalence of risk-alleles differ in ethnic/racial minorities (i.e. SE and GSTM1-null polymorphism), further studies are needed to define the association of smoking and possible gene-smoking interactions and their role in autoimmunity and disease severity in these understudied populations.

ELIGIBILITY:
Inclusion Criteria:

* Meeting ACR criteria for RA

Exclusion Criteria:

* No exclusions

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Omaha VA patients
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2006-10-19 (Actual); Primary Completion 2010-04-01 (Actual); Study Completion 2013-01-01 (Actual)

PRIMARY OUTCOMES:
Rheumatoid factor (RF) antibody status and concentration | baseline
  Rheumatoid factor (RF) antibody status and concentration. RF is an autoantibody that responds to inflammation caused by RA.
Anti-CCP antibody status and concentration | baseline
  Anti-CCP (cyclic citrullinated peptide antibodies) antibody status and concentration.
  The normal level of anti-CCP antibodies is less than 20 units/mL. Anything over this level means a positive test. Anti-cyclic citrullinated peptide antibody titer predicts time to rheumatoid arthritis onset in patients with undifferentiated arthritis.
Evidence of radiographic erosions and scoring. | baseline
  Evidence of radiographic erosions and scoring. Erosions are graded from 0 to 4 (0 = normal; 1 = questionable; 2 = definite but mild; 3 = moderate; and 4 = severe). This method requires a standard reference set of radiographs for comparison. The range of erosion scores is from 0 to 128 in the hands, and from 0 to 48 in the feet.

SECONDARY OUTCOMES:
Smoking status and cotinine levels | baseline
  Smoking status and cotinine levels are recorded. Cotinine is measured in nanograms per milliliter (ng/mL): Cotinine levels in a nonsmoker are generally less than 10 ng/mL. Cotinine levels in a light smoker or someone exposed to secondhand smoke are 11 ng/mL to 30 ng/mL. Cotinine levels in a heavy smoker may be more than 500 ng/mL.
Genotyping of the FSTM1, NAT1, NAT2, and mDEH genes | baseline
  Samples will be taken to genotype FSTM1, NAT1, NAT2, and mDEH genes which are important in carcinogenesis.
Racial/ethnic composition and disease characteristics | baseline
  Both racial/ethnic composition and disease characteristics are recorded for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ted R Mikuls, MD, MSPH, Principal Investigator — University of Nebraska
Locations (1):
- Omaha Veteran's Affairs Medical Center, Omaha, Nebraska, United States

REFERENCES:
- See also: National Institute of Health — http://grants1.nih.gov/grants/oer.htm